CLINICAL TRIAL: NCT06634251
Title: Defining Fluoroscopic Visualization Technique for Optimal Antegrade Entry Point and Anatomical Parameters in Anterior Column Fixation Corridor for Pelvic Surgery: A Novel Perspective
Brief Title: Antegrade Screw Placement Technique in Anterior Column of Acetabulum
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Vedat Öztürk, Specialist Doctor in Orthopedics and Traumatology, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 2024/45-2024-04-01
Record Dates: First submitted 2024-10-08; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Acetabulum Fracture
Keywords: acetabulum fracture; virtual study; anterior column

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- male group: This group consists of 250 healthy male adults whose pelvic CT scans were analyzed to define the optimal antegrade entry point and anatomical parameters for anterior column fixation. The fluoroscopic visualization technique and screw placement were simulated to assess anatomical variations and feasibility specific to the male cohort.
  Interventions: Other: No intervention
- female group: This group consists of 250 healthy female adults whose pelvic CT scans were analyzed to define the optimal antegrade entry point and anatomical parameters for anterior column fixation. The fluoroscopic visualization technique and screw placement were simulated to assess anatomical variations and feasibility specific to the female cohort.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This study is purely observational and does not involve any direct intervention. It utilizes retrospective analysis of computed tomography (CT) scans to simulate the fluoroscopic visualization and screw placement technique in the anterior column fixation corridor (ACFC) of the acetabulum. The objective is to define the optimal antegrade entry point and assess anatomical parameters without performing any physical intervention on the participants.

SUMMARY:
This retrospective observational study aims to define the optimal antegrade entry point for screw placement in the anterior column fixation corridor (ACFC) of the acetabulum. Using fluoroscopic visualization techniques, the study examines computed tomography (CT) scans from 500 healthy adult patients to simulate screw placement and measure anatomical parameters. The goal is to determine patient-specific entry points and to assess the feasibility of screw placement using axial fluoroscopic views. The study also investigates gender-specific anatomical variations to provide insights for safer and more precise screw placement during anterior column fixation in pelvic surgery.

DETAILED DESCRIPTION:
This study focuses on developing and validating a fluoroscopic visualization technique for identifying the optimal antegrade entry point (OAEP) in the anterior column fixation corridor (ACFC) of the acetabulum during pelvic surgery. Using three-dimensional reconstructions from pelvic computed tomography (CT) data of 500 healthy adults, the study simulates screw placement within the ACFC. A cylinder representing the screw is inserted virtually through the OAEP, ensuring that it remains within the confines of the fixation corridor without breaching its boundaries. The study records anatomical measurements, including the corridor's diameter, length, and the angles required for sagittal and coronal plane inclinations to visualize the OAEP.

The study also examines gender-specific anatomical variations, including differences in ACFC diameter, length, and required fluoroscopic angles. By defining patient-specific entry points and establishing a reliable fluoroscopic technique, this study aims to provide a practical and accessible method for anterior column fixation, minimizing complications and improving the safety and precision of screw placement in pelvic surgeries.

This novel approach has the potential to offer a cost-effective alternative to more expensive navigation systems, making it widely applicable in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pelvic computed tomography (CT) scans that provide complete anatomical details of the pelvis.
* Patients aged 18 to 65 years.
* Patients with fully matured bone structures, without evidence of fractures, deformities, or prior orthopedic surgery.
* Patients with no history of rheumatologic disease, advanced osteoporosis, bone metastasis, or metabolic bone disorders.

Exclusion Criteria:

* Patients with pelvic CT scans that do not fully display the anatomical structures.
* Patients younger than 18 years or older than 65 years.
* Patients with pelvic fractures, deformities, or prior orthopedic surgeries.
* Patients with incomplete clinical or radiological data.
* Patients with rheumatologic sequelae, bone metastasis, or metabolic bone diseases.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of 500 healthy adults, including 250 males and 250 females, aged between 18 and 65 years. Participants were selected based on their pelvic computed tomography (CT) scans, which displayed complete and fully matured pelvic anatomy. Individuals with prior orthopedic surgeries, pelvic fractures, deformities, or any bone pathologies such as rheumatologic diseases, advanced osteoporosis, and bone metastasis were excluded. The study focuses on assessing anatomical parameters and optimal entry points for anterior column fixation using fluoroscopic guidance.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Axial Visualization Success | During the simulation of the fluoroscopic imaging, typically within 1 hour of starting the procedure.
  Success in obtaining axial fluoroscopic visualization of the anterior column fixation corridor (ACFC) and optimal antegrade entry point (OAEP).
Screw Placement Feasibility | During the simulation of the screw placement, typically within 1 hour of starting the procedure.
  Feasibility of virtual screw placement within the ACFC without breaching the corridor boundaries.

SECONDARY OUTCOMES:
ACFC Diameter (ACFC-R) | During the simulation of the screw placement, typically within 1 hour of starting the procedure.
  Measurement of the ACFC diameter in millimeters (R) to assess screw placement feasibility.
ACFC Length (ACFC-L) | During the simulation of the screw placement, typically within 1 hour of starting the procedure.
  Measurement of the ACFC length in millimeters (L) to assess screw placement feasibility.
Sagittal Plane Inclination (SPI) | During the simulation of the screw placement, typically within 1 hour of starting the procedure.
  Measurement of the sagittal plane inclination (SPI) required for optimal fluoroscopic visualization of the ACFC.
Coronal Plane Inclination (CPI) | During the simulation of the screw placement, typically within 1 hour of starting the procedure.
  Measurement of the coronal plane inclination (CPI) required for optimal fluoroscopic visualization of the ACFC.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırköy Dr. Sadi Konuk Education and Research Hospital, Department of Orthopedics and Traumatology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided